CLINICAL TRIAL: NCT05829200
Title: Transcranial Doppler(TCD) Evaluation of High Intensity Transient Signals (HITS) in Asymptomatic and Acutely Symptomatic Patients With Carotid Occlusive Disease
Brief Title: Transcranial Doppler(TCD) Evaluation of High Intensity Transient Signals and Carotid Disease
Acronym: TCD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TCD8675309
Record Dates: First submitted 2013-07-08; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Asymptomatic Carotid Stenosis; Symptomatic Carotid Stenosis; TCD; HITS
Keywords: TCD; HITS; Asymptomatic Carotid Stenosis; Symptomatic Carotid Stenosis
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asymptomatic Carotid Disease (Other): All individuals who are consented for elective or urgent carotid endarterectomy would be eligible to participate. If patient gives consent, they would undergo an approximately 30-60 minute Transcranial Doppler (TCD)study. We will collect the number of high intensity transient signals (HITS). The patient would undergo surgery regardless of the TCD result.
  Interventions: Device: Transcranial Doppler (TCD)
- Symtomatic Carotid Disease (Other): All individuals who are consented for elective or urgent carotid endarterectomy would be eligible to participate. If patient gives consent, they would undergo an approximately 30-60 minute Transcranial Doppler (TCD)study. We will collect the number of high intensity transient signals (HITS). The patient would undergo surgery regardless of the TCD result.
  Interventions: Device: Transcranial Doppler (TCD)

INTERVENTIONS:
Device: Transcranial Doppler (TCD) — All individuals who are consented for elective or urgent carotid endarterectomy would be eligible to participate. If patient gives consent, they would undergo an approximately 30-60 minute TCD study. We will collect the number of high intensity transient signals (HITS). The patient would undergo surgery regardless of the TCD result.

SUMMARY:
Carotid Disease causes 10% of strokes. The Investigators are attempting to investigate the use of Transcranial Doppler to see if this is and effective, efficient, and/or valid way to identify individuals at highest risk for thromboembolic events from carotid disease. The plan is to plot the number of high intensity transient transcranial doppler signals with the category of patient (asymptomatic, symptomatic, and actively symptomatic) and evaluate if a relationship exists. The Investigators hypothesize that a linear relationship exists in that the higher the number of HITS the more symptomatic the patient. If results demonstrate the numbers of HITS correlate with the severity of disease this could potentially identify asymptomatic patients having subclinical symptoms who would benefit from a more urgent surgical intervention versus the current standard of care of elective intervention.

DETAILED DESCRIPTION:
Approximately 20% of strokes are attributable to carotid stenosis through atheroembolic events. Ischemic stroke confers a significant morbidity and mortality. Operative intervention (carotid endarterectomy [CEA]) has proven to decrease the risk of ischemic stroke. The guidelines for patient selection for carotid surgical intervention were established in the 1990s and have proven reasonably adequate, however with improving technology there may be modalities that can identify patients that may be at a higher risk than initially thought. One such modality that is under investigation is the use of transcranial doppler (TCD).

Presently, TCD is primarily used in conjunction with neuro-interventionalist related procedures (cerebral angiogram/stenting/coiling) to monitor for vasospasm and blood flow within the cerebral circulation. The technology assessment report of the American Academy of Neurology published in 1990 stated that TCD has established value in the assessment of patients with intracranial stenosis, collaterals, subarachnoid hemorrhage, and brain death. TCD has been used during intraoperative carotid endarterectomy to evaluate blood flow and need for arterial shunting. Recently, it has been used to identify and detect microemboli via the evaluation of high intensity transient signals (HITS). It has been shown in asymptomatic carotid patients that aggressive medical management can decrease the number of HITS on TCD potentially conferring a decrease in stroke. There is more literature evolving that demonstrates the potential of TCD being used to assist in patient selection for surgical intervention (carotid endarterectomy); however the studies have not yet been conducted. Our study is the first step in beginning this process.

The current standard of care is to consider surgical intervention for the following three groups of patients with carotid stenosis (a narrowing of the internal carotid artery): asymptomatic patients are defined as patients who have not experienced a transient ischemic attack (TIA) and/or stroke-like symptoms who have been identified as having a high grade carotid stenosis (narrowing of the internal carotid artery of greater than 80% via CTA, Carotid Doppler Ultrasound, and/or MRA); symptomatic patients who have previously experienced a ischemic stroke or TIA (no active symptoms at the time of presentation) and have 50% or greater carotid stenosis diagnosed by the same imaging modalities; the third group are individuals who present to the hospital as their ischemic symptoms have recently or are actively occurring with 50% or greater stenosis, unfavorable plaque, and/or acute carotid occlusion (diagnosed by the same imaging modalities). Our study proposes that the aforementioned patients undergo TCD to evaluate the number of HITS prior to surgical intervention.

TCD is a non-invasive study. It does not involve injection of any contrast material or the need for blood work prior to its undertaking. The test itself takes 30-60 minutes. The test would be administered by one specifically trained ultrasound technician. The TCD information will not affect patient care in any way; no definitive treatment will be delayed. The number of HITS would not change the type or timing of surgical intervention.

This is a prospective study. The first two groups of patients are generally referred to Ochsner's vascular surgeons and if eligible for surgical intervention during a clinic visit would be electively referred to get the non-invasive TCD test. There are some individuals in the second group who may have been admitted to the hospital and their symptoms have resolved. This group would be identified by neurology and radiology members of the stroke team via consult to the vascular surgery service. The TCD could be done while the patient was hospitalized. The third group is identified during a stroke code process. If the patient is found to meet surgical criteria the patient would undergo TCD in the emergency department or on the floors upon admission. The TCD order would be initiated by the stroke code team or vascular surgery.

The TCD reports would be forwarded to and kept by the study coordinator.

The plan would then be to plot the number of HITS with the category of patient (asymptomatic, symptomatic, and actively symptomatic) and evaluate if a relationship exists. The Investigators hypothesize that a linear relationship exists in that the higher the number of HITS the more symptomatic the patient. If results demonstrate the numbers of HITS correlate with the severity of disease this could potentially identify asymptomatic patients having subclinical symptoms who would benefit from a more urgent surgical intervention versus the current standard of care of elective intervention.

ELIGIBILITY:
Inclusion Criteria:

• Any individual consented for elective or urgent carotid endarterectomy (asymptomatic stenosis >80% and/or symptomatic carotid stenosis >50%).

Exclusion Criteria:

* Any individual who is unstable and needs to go to the operating room emergently is excluded from this study.
* Any individual who can not tolerate a TCD exam will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of HITS | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hernan Bazan, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States